CLINICAL TRIAL: NCT05057572
Title: Efficacy and Safety of Carvedilol in Cirrhosis Patients With Uncomplicated Ascites Without High Risk Esophageal Varices- A Randomised Controlled Trial"
Brief Title: Efficacy and Safety of Carvedilol in Cirrhosis Patients With Uncomplicated Ascites Without High Risk Esophageal Varices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-44
Record Dates: First submitted 2021-09-08; First posted 2021-09-27 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carvedilol with Standard Medical Treatment (Experimental): Arm A will receive carvedilol plus standard medical therpy,Carvedilol: will be started with initial dose of 3.125 mg BD then After 3 days, increase the dose to 6.25 mg BD, Maximum dose would be 12.5 mg BD, the same shall be switch to Maximum tollrated dose if SBP >90, HR >55.
  Interventions: Drug: Carvedilol; Drug: Standard Medical Treatment
- Standard Medical Treatment (Active Comparator): - Arm B will receive standard medical therapy.SMT (as described) that is Grade II ascites - Lasilactone (20/50) OD then Change after 1 week as per response, monitor diuretic intolerance.
  Interventions: Drug: Standard Medical Treatment

INTERVENTIONS:
Drug: Carvedilol — - Arm A will receive carvedilol plus standard medical therpy,Carvedilol: will be started with initial dose of 3.125 mg BD then After 3 days, increase the dose to 6.25 mg BD, Maximum dose would be 12.5 mg BD, the same shall be switch to Maximum tollrated dose if SBP>90, HR >55.
  Arms: Carvedilol with Standard Medical Treatment
Drug: Standard Medical Treatment — * Arm B will receive standard medical therapy.SMT (as described) that is Grade II ascites - Lasilactone (20/50) OD then Change after 1 week as per response, monitor diuretic intolerance.
  * Grade III ascites will undergo large volume paracentesis, lasilactone (20/50) OD Both groups will receive albumin as indicated (LT references as per protocol will be send for eligible patients)

SUMMARY:
The cumulative risk of refractory ascites is in the order of 20% within five years of the development of ascites. An elevated sinusoidal pressure is essential for the development of ascites, as fluid accumulation does not develop at portal pressure gradient below 8 mm Hg, and rising corrected sinusoidal pressure correlates with decreased 24-hour urinary excretion of sodium.More recently, it has been hypothesised that bacterial translocation associated with portal hypertension in cirrhosis and related pathogen-associated, molecular pattern activated innate immune responses lead to systemic inflammation.This is associated with vasodilatation as well as release of proinflammatory cytokines, reactive oxygen and nitrogen species, contributing to organ dysfunction.This activates sympathetic nervous system stimulating reabsorption of sodium in proximal,distal tubules, loop of Henle and collecting duct as well as the renin-angiotensin-aldosterone system, leading to sodium absorption from distal tubule and collecting duct.[5]Renal sodium retention and eventual free water clearance due to non-osmoticrelease of arginine-vasopressin and its action on V2 receptor in the collectingduct underlie the fluid retention associated with oedema and ascites in cirrhosis.The lowering of portal pressure using non selective beta blocker has also been shown to reduce the development of ascites, refractory ascites and hepatorenal syndrome.Furthermore, the effect of non slective beta blocker on intestinal permeability, bacterial translocation and inflammatory response has been proposed to mitigate the risk of developing spontaneous bacterial peritonitis.

DETAILED DESCRIPTION:
AIM-To compare the safety and efficacy of addition of carvedilol to SMT (diuretics +/- albumin) compared to SMT alone in the prevention of complicated ascites (refractory ascites, AKI-HRS, SBP or severe hyponatremia) at 1year.

Methodology:

Study population: Patient of liver cirrhosis presenting with uncomplicated ascites and without high risk esophageal varices.

Study design:

* A prospective, randomized, single center open label study.
* The study will be conducted on the consecutive patients presenting with uncomplicated ascites and low risk esophageal varices seen at the outpatient clinics/wards of Department of Hepatology, ILBS, New Delhi from July 2021 to June 2023.

Study period: 2years from the date of ethics approval

Sample size with justification:

* Assuming that the complication rate in carvedilol group is 8% and placebo 30% so the complication free rate of 92% and 70 % further assuming alpha -5%, power 80%.
* Investigator need to enrol 108 cases in two groups further with 10% drop out rate it was decided to enroll 120 cases
* Randomisation into two groups by block randomisation method,taking block size 8

Intervention:

* Patients will be randomized into two Arms A & B.
* Arm A will receive carvedilol plus standard medical therpy,Carvedilol: will be started with initial dose of 3.125 mg BD then After 3 days, increase the dose to 6.25 mg BD, Maximum dose would be 12.5 mg BD, the same shall be switch to Maximum tollrated dose if SBP >90, HR >55.
* Arm B will receive standard medical therapy.SMT (as described) that is
* Grade II ascites - Lasilactone (20/50) OD then Change after 1 week as per response, monitor diuretic intolerance.
* Grade III ascites will undergo large volume paracentesis, lasilactone (20/50) OD Both groups will receive albumin as indicated (LT references as per protocol will be send for eligible patients)
* For Diuretic intolerance -Na, K, urea, creatnine will be monitred first weekly then once monthly then SOS as per need
* For Carvedilol heart rate will be monitored first weekly then monthly then SOS as per need
* Dose of carvedilol will be adjusted as per protocol.
* Other treatments given: Alumbin infusion to both group, lasilactone.
* Complications / Organ failures (3m, 6m, 1y or detected during tele/online consult or on opd basis
* Data to be collected

  * Baseline -
  * Blood : KFT, LFT, CBC, INR, IL-6, CRP,TNF Alpha
  * Imaging : USG upper abdomen and doppler for renal blood flow,
  * 2D ECHO
  * Urine : Urine R/E, Urine Na,AFP
  * A/F analysis - for SBP
  * HVPG, UGIE
  * At 3 months, 6 months.
  * Blood : LFT, KFT, INR,AFP
  * At 1 year
  * Blood : KFT, LFT, CBC, INR, TNF alpha,IL-6, CRP,AFP
  * Imaging : USG upper abdomen
  * Urine : Urine Na
  * HVPG, UGIE

Statistical Analysis:

Data will be reported as mean + SD. Categorical variables will be compared using the chi-square test or Fisher exact test. Normal continuous variables will be compared using the Student's t testNon normal continuous variables will be compared using the Mann Whitney rank-sum test (unpaired data) or the Wilcoxon test (paired data). The actuarial probability of survival will be calculated by the Kaplan-Meier method and compared using the log-rank test.A Cox regression analysis will be performed to identify independent prognostic factors for survival.Univariate and multivariate analysis will be used whenever applicable.

Adverse effects:

Hypotension (2.6-17.6%) with minor side effets as fainting, shortness of breath, weight gain, swelling of the arms, hands, feet, ankles, or lower legs, chest pain, slow or irregular heartbeat, rash, itching, difficulty breathing and swallowing tiredness, weakness, lightheadedness, dizziness, headache, diarrhea, nausea, vomiting, vision change, joint pain difficulty falling asleep or staying asleep, cough dry eyes, numbness, burning, or tingling in the arms or legs.

Stopping rule of study:

* Severe complications requiring discontinuation of therapy severe Respiratory distress, severe bradycardia heart block not responding to dose reduction.
* Patient refusal to further participate in study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Liver cirrhosis
* Grade II-III high SAAG ascites
* Small low risk or no esophageal varices
* CTP 7-12

Exclusion Criteria:

* Age <18 years
* AKI at enrollement (Prior transient volume responsive AKI stage I included)
* Post renal or liver transplantation
* History of CAD, PVD, ventricular arrythmia, Bronchial asthma
* SBP at diagnosis
* Severe Hyponatremia (Na <125 MEq/L)
* Grade II/III/IV HE
* Advanced HCC (BCLC C,D), PVTT, Pregnancy or Lactating mother
* High risk varices (Large varices or small high risk varices)
* CTP >12
* ACLF
* Mixed / TB ascites
* Bilirubin >5 mg/dl
* Known CKD, obstructive uropathy
* Patient on MV, NIV, systemic sepsis and shock
* Lack of informed consent
* Prior intolerance or S/E to carvedilol or diuretics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Complicated ascites (any of refractory ascites, SBP, AKI-HRS) | 1 year

SECONDARY OUTCOMES:
Ascites resolution in both groups | 3 Months
  Ascites well controlled with appropriate medical treatment, i.e, the minimum diuretic dose necessary to control weight gain and ascites formation that did not lead to diuretic-induced complications, such as renal impairment, hyponatremia, hypokalemia or hyperkalemia, or HE
Ascites resolution in both groups | 6 Months
  Ascites well controlled with appropriate medical treatment, i.e, the minimum diuretic dose necessary to control weight gain and ascites formation that did not lead to diuretic-induced complications, such as renal impairment, hyponatremia, hypokalemia or hyperkalemia, or HE
Ascites resolution in both groups | 1 year
  Ascites well controlled with appropriate medical treatment, i.e, the minimum diuretic dose necessary to control weight gain and ascites formation that did not lead to diuretic-induced complications, such as renal impairment, hyponatremia, hypokalemia or hyperkalemia, or HE
Need and frequency of Large Volume Paracentesis | 1 year
Incidence of PICD in 1 year | 1 year
Mortality | 1 year
Change in grade of varices in both groups | 1 year
  Change is defined as from garde I to garde II/ grade III
Reduction in HVPG in both groups | 1 year
Change in MELD score in both groups | 3 months
  Minimum MELD=6 Maximum MELD=40
Change in MELD score in both groups | 6 months
  Minimum MELD=6 Maximum MELD=40
Change in MELD score in both groups | 1 year
  Minimum MELD=6 Maximum MELD=40
Change in CTP score in both groups | 3 months
  CTP Change is CTP- C to CTP- B & CTP- B to CTP- A
Change in CTP score in both groups | 6 months
  CTP Change is CTP- C to CTP- B & CTP- B to CTP- A
Change in CTP score in both groups | 1 year
  CTP Change is CTP- C to CTP- B & CTP- B to CTP- A
Incidence of HE in both groups | 6 months
Incidence of HE in both groups. | 1 year
Incidence of variceal bleed in both groups | 6 months
Incidence of variceal bleed in both groups | 1 year
Incidence of AKI in both groups | 6 months
Incidence of AKI in both groups | 1 year
Incidence of SBP in both groups | 6 months
Incidence of SBP in both groups | 1 year
Incidence of severe hyponatremia in both groups | 6 months
Incidence of severe hyponatremia in both groups | 1 year
Incidence of refractory ascites in both groups | 6 months
Incidence of refractory ascites in both groups | 1 year
Maximum tolerated dose of carvedilol | 1 year
Tretament (carvedilol) related adverse events and their grades | 1 year
  Adverse Events are defined as incidence of Bradycardia,Hypotension,Breathlessness

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Khajuria R, Jindal A, Sharma MK, Arora V, Vyas AK, Kumar G, Sarin SK. Efficacy and Safety of Carvedilol in Cirrhosis Patients With New-Onset Uncomplicated Ascites Without High-Risk Esophageal Varices (CARVE-AS Trial). Am J Gastroenterol. 2025 Jul 21. doi: 10.14309/ajg.0000000000003650. Online ahead of print. PMID 40689908